CLINICAL TRIAL: NCT02723734
Title: A Validation Study on the Impact of Decipher® Testing on Treatment Recommendations in African-American and Non-African American Men With Prostate Cancer (VANDAAM Study)
Brief Title: Validation Study on the Impact of Decipher® Testing - VANDAAM Study
Acronym: VANDAAM
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-18523
Record Dates: First submitted 2016-03-15; First posted 2016-03-30 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Decipher®; African-American men; prostate; low risk PCa; intermediate risk PCa; genomic classifier (GC)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One PCa biopsy specimen (collected at baseline for all participants). One PCa RP specimen (only for those participants that select surgery). Blood Specimen (collected at baseline for all participants if they agree to participate in blood draw).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African-American Men (AAM): AAM with low risk or intermediate risk prostate cancer (PCa). Decipher® testing and standard treatment.
  Interventions: Other: Decipher® Testing
- Non-African American Men (NAAM): NAAM with low risk or intermediate risk prostate cancer (PCa). Decipher® testing and standard treatment.
  Interventions: Other: Decipher® Testing

INTERVENTIONS:
Other: Decipher® Testing — Decipher® Prostate Cancer Classifier (Post-Op and Biopsy), a Genomic Classifier (GC) test. Biopsy and prostatectomy specimens will be collected for GC testing.
  Other Names: Genomic Classifier (GC) test

SUMMARY:
The primary purpose of this study is to determine whether a tumor test recently developed by GenomeDx Biosciences known as Decipher® can predict aggressive prostate cancer with the same accuracy in African-American men (AAM) as in non-African-American men (NAAM). The Decipher® test was developed from samples derived mainly from men of European origins and little is known about its performance in AAM. It is important to study whether this test can be used in AAM who are known to experience the highest rates of prostate cancer as well as death from prostate cancer. The use of the Decipher® test result to predict how well a patient will do before treatment may make it possible for doctors to distinguish aggressive disease from low risk prostate cancer and modify treatment accordingly. Thus, patients that do not need additional therapies may be spared from unnecessary side effects and those that are at risk may be provided with more aggressive therapy to improve survival. This study is being done to learn whether the Decipher test can really affect these outcomes.

DETAILED DESCRIPTION:
This is a multisite, prospective validation trial. Based on a population consisting of 25% AAM and 75% NAAM, investigators will actively recruit participants and aim to achieve a 1:1 enrollment ratio of AAM to NAAM. To achieve this, low risk AAM will be accrued first and then matching NAAM will be enrolled. NAAM men will be matched to AAM on prostate specific antigen (PSA) at diagnosis.

There will be no treatment intervention beyond standard of care (SOC), and therefore participants will be allowed to choose their definitive treatment option. The intent is to enroll low risk and high volume disease (burden) patients to limit the accrual of patients that would select active surveillance (AS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Karnofsky Performance Status >70
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Pathologically (histologically) proven diagnosis of prostate cancer (PCa) undergoing their first line of treatment
* Meet National Comprehensive Cancer Network (NCCN) criteria for either: Low risk PCa (defined as Gleason score 6 in ≥ 3 cores; T-stage T1c- T2a); Intermediate risk PCa (defined as Gleason score 7, or prostatic specific antigen (PSA) ≥ 10 ng/ml & < 20 ng/ml, or T-stage ≤ T2c)
* Eligible for either radical prostatectomy (RP) or definitive radiation therapy (RT) (+/- short-term androgen deprivation therapy (ADT))
* Age > 18 years
* Biopsy specimen available

Exclusion Criteria:

* Inability to acquire biopsy or prostatectomy tissue
* History of prior PCa directed chemotherapy or pelvic irradiation (prior to study enrollment)
* Documented distant metastatic disease or pelvic lymphadenopathy
* Prior radical prostatectomy (RP) or cryosurgery for prostate cancer or bilateral orchiectomy
* Targeted for active surveillance after diagnostic biopsy
* Selecting ADT alone after diagnostic biopsy
* On active surveillance for > 6 months after diagnosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Two Year Prostatic Specific Antigen (PSA) Failure Rate | Up to 24 months
  PSA failure defined for first line treatment options of Radical Prostatectomy (RP) and Radiotherapy (RT) in accordance with National Comprehensive Cancer Network (NCCN) guidelines: PSA failure for RP is defined by an undetectable PSA after surgery with a subsequent detectable PSA that increases on 2 or more determinations (PSA recurrence); or failure of PSA to fall to undetectable levels (PSA persistence). PSA failure for treatment with RT is defined as PSA increase by 2 ng/mL or more above the nadir PSA.
  To estimate the performance of genomic classifier (GC) in predicting 2-yr PSA failure rate, the area under curve (AUC) of a standard Receiver Operating Characteristic (ROC) curve will be calculated with corresponding 95% confidence intervals using resampling methods. In addition, positive and negative predictive probabilities, sensitivity, specificity and accuracy and associated 95% confidence intervals will also be calculated using predefined cut-points of 0.45 and 0.60.

CONTACTS AND LOCATIONS:
Overall Officials: Kosj Yamoah, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - Bay Pines VA Health care System, Bay Pines, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - James A. Haley VA Hospital, Tampa, Florida

REFERENCES:
- [Result] Awasthi S, Grass GD, Torres-Roca J, Johnstone PAS, Pow-Sang J, Dhillon J, Park J, Rounbehler RJ, Davicioni E, Hakansson A, Liu Y, Fink AK, DeRenzis A, Creed JH, Poch M, Li R, Manley B, Fernandez D, Naghavi A, Gage K, Lu-Yao G, Katsoulakis E, Burri RJ, Leone A, Ercole CE, Palmer JD, Vapiwala N, Deville C, Rebbeck TR, Dicker AP, Kelly W, Yamoah K. Genomic Testing in Localized Prostate Cancer Can Identify Subsets of African Americans With Aggressive Disease. J Natl Cancer Inst. 2022 Dec 8;114(12):1656-1664. doi: 10.1093/jnci/djac162. PMID 36053178
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/